CLINICAL TRIAL: NCT00230893
Title: Characterization of the Use of Antipsychotics in PTSD During the Past Seven Years
Status: Completed | Type: Observational
Sponsor: Tuscaloosa Research & Education Advancement Corporation (Other)
Collaborators: Janssen, LP (Industry)
Other Study IDs: TREAC - PTSD Retrospective; TREAC - PTSD Retrospective
Record Dates: First submitted 2005-09-29; First posted 2005-10-03 (Estimated); Last update posted 2006-09-21 (Estimated); Status verified 2006-09

CONDITIONS: PTSD; Post-Traumatic Stress Disorder
Keywords: Antipsychotics; PTSD; Post Traumatic Stress Disorder; monotherapy; adjunct therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Retrospective

SUMMARY:
The primary objective is to examine the percentage of patients with PTSD who were prescribed an antipsychotic over the past seven years in the VA Network 7 (AL, GA, SC) and compare the percentage on an annual basis. We will also determine the type and dose of antipsychotics received. We hypothesize that there has been a significant increase in antipsychotic use, especially atypical antipsychotics, prescribed for patients with PTSD over the last 7 years

DETAILED DESCRIPTION:
This study is a retrospective electronic review of the VISN 7 Data Warehouse to determine what have been the emerging trends in prescriptions of atypical antipsychotic medications over the past seven years for the treatment of posttraumatic stress disorder (PTSD) in the VA

This study is a retrospective electronic review of patients of the VISN 7 Data Warehouse of patients with a diagnosis of PTSD treated with antipsychotics as monotherapy or adjunctive therapy at a VA Medical Center or VA clinic in VISN 7 (GA, SC, and AL). The data will be retrieved from a computerized list of patients treated in VA VISN 7 for PTSD from 1998-2005 and cross-referenced with the electronic pharmacy file for having received a prescription of an antipsychotic medication. No personal identifiers will be collected. The data will then be examined to determine what type of antipsychotics were prescribed and the dose and duration of the antipsychotics. In addition, demographics and clinical characteristics available through the Data Warehouse will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, any race or ethnic origin at least 19 years of age.
* Patients with a diagnosis of PTSD
* Treated with an antipsychotic as a monotherapy or adjunctive therapy
* Patient must have been seen at a VA medical center or clinic within VISN 7 during the study period.

Exclusion Criteria:

* Patients not diagnosed with PTSD
* Not treated with an antipsychotic as a monotherapy or adjunctive therapy
* Patients outside of Network 7
* Patients with a diagnosis of schizophrenia, schizoaffective disorder, or bipolar disorder

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99
Dates: Start 2005-07; Study Completion 2005-09

CONTACTS AND LOCATIONS:
Overall Officials: Lori L. Davis, MD, Principal Investigator — Tuscaloosa Veterans Affairs Medical Center
Locations (1):
- Tuscaloosa VA Medical Center, Tuscaloosa, Alabama, United States

REFERENCES:
- [Background] Kozaric-Kovacic D, Pivac N, Muck-Seler D, Rothbaum BO. Risperidone in psychotic combat-related posttraumatic stress disorder: an open trial. J Clin Psychiatry. 2005 Jul;66(7):922-7. doi: 10.4088/jcp.v66n0716. PMID 16013909